CLINICAL TRIAL: NCT04078711
Title: Qianyangyuyin Formula Prevent and Treat for Early Renal Injury in Hypertensive Patients
Brief Title: Chinese Medicine Treat for Hypertensive Renal Injury
Acronym: CHAIR
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhu-Yuan Fang, Professor, Jiangsu Province Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019NL-086-02
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Hypertension; Renal Injury
Keywords: hypertension; chronic kidney disease; traditional chinese medicine; early renal injury; albumin to creatinine ratio(UACR)
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- losartan & qianyangyuyin (Experimental): Losartan 100mg tablet (if necessary combined with CCBs) by mouth, qd for 6 months and Chinese Medicine (Qianyangyuyin granule) 20g by mouth, bid for 6 months.
  Interventions: Drug: Losartan 100Mg Tab; Drug: Qianyangyuyin 20g Granule
- Losartan & Placebo (Placebo Comparator): Losartan 100mg tablet (if necessary combined with CCBs) by mouth, qd for 6 months and Qianyangyuyin placebo 20g by mouth, bid for 6 months.
  Interventions: Drug: Losartan 100Mg Tab; Drug: placebo

INTERVENTIONS:
Drug: Losartan 100Mg Tab — 100Mg Tab, qd, po, 6 months
  Other Names: Cozaar
Drug: Qianyangyuyin 20g Granule — 20g, Granule, bid, po, 6 months
  Arms: losartan & qianyangyuyin
Drug: placebo — Similar granule manufactured to mimic qianyangyuyin granule, 20g, Granule, bid, po, 6 months
  Other Names: placebo(qianyangyuyin)
  Arms: Losartan & Placebo

SUMMARY:
This study evaluates whether the traditional chinese medicine (Qianyangyuyin formula) could prevent and treat early renal injury in patients with hypertension and microalbuminuria (defined as a urinary albumin to creatinine ratio between 30 and 300 mg/g) based on standard antihypertensive treatment.

DETAILED DESCRIPTION:
Hypertension is the main cardiovascular disease and the most important risk factor for severe lethal and disabling diseases such as stroke, myocardial infarction, heart failure, and chronic renal insufficiency. The higher the blood pressure level, the higher the risk of these diseases. Antihypertensive drugs can control blood pressure, and effectively reduce the risk of these serious complications. A multi-center, randomized, parallel, placebo-controlled clinical study was designed to explore the effectiveness and safety of early intervention of Chinese medicine (Qianyanguuyin formula) in improving urinary albumin to creatinine ratio (ACR), based on standard antihypertensive treatment (losartan 100mg qd, if necessary combined with calcium channel blockers). Patients were recruited if they were (1) age between 35 and 55 years old, (2) primary hypertension (grades 2-3 ), (3) microalbuminuria (ACR of 30-300 mg/g) and eGFR of at least 60 ml / (min∙1.73m2), (4) ascendant hyperactivity of liver Yang or Yin deficiency in TCM syndrome. It's intented to form a standardized plan for the prevention and treatment of early renal injury in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has primary hypertension(grades 2-3)
* Subject has microalbuminuria [defined as a urinary albumin/creatinine ratio (UACR) between 30 and 300mg/g, and a eGFR at least 60ml/(min∙1.73m2)]
* Subject has ascendant hyperactivity of liver Yang or Yin deficiency in TCM syndrome
* Subject voluntarily participates in the trial and signs informed consent

Exclusion Criteria:

* Subject has secondary hypertension
* Subject with pregnancy or lactating
* Subject has serious life-threatening diseases, such as acute myocardial infarction, stroke, heart failure (NYHA IV), and malignant arrhythmia
* Subject's liver function (AST or ALT) is 2 times greater than normal value
* Subject has history of mental illness
* Subject currently participates in other drug clinical trials

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
albumin-to-creatinine ratio(UACR) | 6 months
  UACR tested at baseline and each month. Microalbuminuria was defined as urinary ACR of at least 30mg/g.

SECONDARY OUTCOMES:
Ambulatory blood pressure level | 6 months
  ABPM was measured at baseline, 3 and 6 months. Both systolic and diastolic pressure was assessed. Hypertension was defined as mean ambulatory blood pressure of at least 130/80 mmHg.
Office blood pressure level 6/5000 Office blood pressure level | 6 months
  Office blood pressure was measured at baseline and each month. Both systolic and diastolic pressure was assessed. Hypertension was defined as office blood pressure of at least 140/90 mmHg.
Traditional Chinese Medicine syndrome scores | 6 months
  Self reported TCM syndrome scores at baseline and each month. Each main symptom is scored 0、2、4、6 (0 = no sympton; 6 = as heavy as can be), and each secondary symptom is scored 0、1、2、3(0=no symptom; 3= as heavy as can be).

CONTACTS AND LOCATIONS:
Overall Officials: Zhuyuan Fang, Principal Investigator — Jiangsu Province Hospital of Traditional Chinese Medicine; Ming Liu, Study Director — Jiangsu Province Hospital of Traditional Chinese Medicine

REFERENCES:
- [Background] Gaziano TA, Bitton A, Anand S, Weinstein MC; International Society of Hypertension. The global cost of nonoptimal blood pressure. J Hypertens. 2009 Jul;27(7):1472-7. doi: 10.1097/HJH.0b013e32832a9ba3. PMID 19474763
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Kunz R, Friedrich C, Wolbers M, Mann JF. Meta-analysis: effect of monotherapy and combination therapy with inhibitors of the renin angiotensin system on proteinuria in renal disease. Ann Intern Med. 2008 Jan 1;148(1):30-48. doi: 10.7326/0003-4819-148-1-200801010-00190. Epub 2007 Nov 5. PMID 17984482
- [Background] Haller H, Ito S, Izzo JL Jr, Januszewicz A, Katayama S, Menne J, Mimran A, Rabelink TJ, Ritz E, Ruilope LM, Rump LC, Viberti G; ROADMAP Trial Investigators. Olmesartan for the delay or prevention of microalbuminuria in type 2 diabetes. N Engl J Med. 2011 Mar 10;364(10):907-17. doi: 10.1056/NEJMoa1007994. PMID 21388309
- [Background] Ruggenenti P, Fassi A, Ilieva A, Iliev IP, Chiurchiu C, Rubis N, Gherardi G, Ene-Iordache B, Gaspari F, Perna A, Cravedi P, Bossi A, Trevisan R, Motterlini N, Remuzzi G; BENEDICT-B Study Investigators. Effects of verapamil added-on trandolapril therapy in hypertensive type 2 diabetes patients with microalbuminuria: the BENEDICT-B randomized trial. J Hypertens. 2011 Feb;29(2):207-16. doi: 10.1097/hjh.0b013e32834069bd. PMID 21243736
- [Background] Li X, Zhang J, Huang J, Ma A, Yang J, Li W, Wu Z, Yao C, Zhang Y, Yao W, Zhang B, Gao R; Efficacy and Safety of Qili Qiangxin Capsules for Chronic Heart Failure Study Group. A multicenter, randomized, double-blind, parallel-group, placebo-controlled study of the effects of qili qiangxin capsules in patients with chronic heart failure. J Am Coll Cardiol. 2013 Sep 17;62(12):1065-1072. doi: 10.1016/j.jacc.2013.05.035. Epub 2013 Jun 7. PMID 23747768
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Joint Committee for Guideline Revision. 2018 Chinese Guidelines for Prevention and Treatment of Hypertension-A report of the Revision Committee of Chinese Guidelines for Prevention and Treatment of Hypertension. J Geriatr Cardiol. 2019 Mar;16(3):182-241. doi: 10.11909/j.issn.1671-5411.2019.03.014. No abstract available. PMID 31080465
- [Background] Schmieder RE, Hilgers KF, Schlaich MP, Schmidt BM. Renin-angiotensin system and cardiovascular risk. Lancet. 2007 Apr 7;369(9568):1208-19. doi: 10.1016/S0140-6736(07)60242-6. PMID 17416265

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT04078711/Prot_SAP_000.pdf